CLINICAL TRIAL: NCT00088556
Title: Phase 1-2a Dose-Ranging Study of the Triplet Combination of Carboplatin, Paclitaxel and TLK286 as First-Line Therapy in Advanced Non-Small Cell Lung Cancer
Brief Title: Carboplatin, Paclitaxel and TLK286 (Telcyta) as First-Line Therapy in Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Telik (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TLK286.2023
Record Dates: First submitted 2004-07-29; First posted 2004-07-30 (Estimated); Last update posted 2012-05-31 (Estimated); Status verified 2011-06

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — TER 286; Carboplatin; Paclitaxel

ARMS (1):
- Triplet Combination of TLK286 Carboplatin & Paclitaxel (Experimental): Experimental
  Interventions: Drug: TLK286; Drug: carboplatin; Drug: paclitaxel

INTERVENTIONS:
Drug: TLK286 — Every 3 Weeks with a starting dose of TLK286 @ 400 mg/m²
Drug: carboplatin — AUC 6 mg/mL/min Once every 3 weeks
Drug: paclitaxel — 200 mg/m² Once every 3 weeks

SUMMARY:
The purpose of this trial is to study the efficacy and safety of the triplet combination of TLK286, carboplatin and paclitaxel as first-line therapy for patients with advanced non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Histologically confirmed non-small cell lung cancer (NSCLC)
* Stage IV or IIIB (disease that is not eligible for combined modality chemotherapy and radiation)
* Measurable disease by RECIST
* ECOG status of 0-1
* Adequate liver and renal function
* Adequate bone marrow reserves

Exclusion Criteria:

* Prior chemotherapy, immunotherapy or biologic therapy for metastatic NSCLC
* Up to one prior adjuvant or neoadjuvant chemotherapy is allowed
* History of bone marrow transplantation or stem cell support
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2004-08; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Study Objectives | Every 6 Weeks
  1. To determine the MTD of patients treated with the triplet combination of TLK286, paclitaxel and carboplatin
  2. To determine the safety of patients treated with the triplet combination of TLK286, paclitaxel and carboplatin
  3. To determine the objective response rate (ORR) of patients treated with the triplet combination of TLK286, paclitaxel and carboplatin

CONTACTS AND LOCATIONS:
Locations (47):
- United States (47):
  - Bay Area Cancer Research Group, Concord, California
  - East Bay Medical Oncology/Hematology Associates, Concord, California
  - Southwest Cancer Care, Escondido, California
  - Kaiser Permanente Medical Center, Hayward, California
  - Southwest Cancer Care, Murrieta, California
  - Kaiser Permanente Medical Center, Oakland, California
  - Southwest Cancer Care, Poway, California
  - Kaiser Permanente Medical Center, Sacramento, California
  - Kaiser Permanente Medical Center, San Francisco, California
  - Kaiser Permanente Medical Center, San Jose, California
  - Kaiser Permanente Medical Center, Santa Clara, California
  - Kaiser Permanente Medical Center, So. San Francisco, California
  - Kaiser Permanente Medical Center, Vallejo, California
  - Diablo Valley Oncology & Hematology Medical Group, Walnut Creek, California
  - Kaiser Permanente Medical Center, Walnut Creek, California
  - Citrus Hematology and Oncology, Crystal River, Florida
  - Citrus Hematology and Oncology Center, Inverness, Florida
  - Florida Wellcare Alliance, LC, Inverness, Florida
  - Kansas City Cancer Center, Kansas City, Kansas
  - Kansas City Cancer Center - Central Research Dept. Data Office & Drug Discovery Location, Lenexa, Kansas
  - Kansas City Cancer Center, Overland Park, Kansas
  - Department of Veterns Affairs - Overton Brooks VA Medical Center, Shreveport, Louisiana
  - LSU Health Sciences Center, Shreveport, Louisiana
  - University of Maryland, Baltimore University of Maryland Medical System-Greenebaum Cancer Center, Baltimore, Maryland
  - Center for Cancer and Blood Disorders, P. C., Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Kansas City Cancer Center, Kansas City, Missouri
  - Kansas City Cancer Center, Lee's Summit, Missouri
  - St. John's Mercy Medical Center, St Louis, Missouri
  - St. John's Mercy Hospital, Washington, Missouri
  - Clinical Research Service, Scottsbluff, Nebraska
  - Horizons West Medical Group, Scottsbluff, Nebraska
  - Dakota Cancer Institute, Fargo, North Dakota
  - Odyssey Research, Fargo, North Dakota
  - Tennessee Oncology, PLLC, Clarksville, Tennessee
  - Tennessee Oncology, PLLC, Franklin, Tennessee
  - Tennessee Oncology, PLLC, Hermitage, Tennessee
  - Tennessee Oncology, PLLC, Lebanon, Tennessee
  - Tennessee Oncology, PLLC, Murfreesboro, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Tennessee Oncology, PLLC, Smyrna, Tennessee
  - Texas Cancer Associates, Dallas, Texas
  - Texas Cancer Associates, Plano, Texas
  - Danville Hematology & Oncology, Inc., Danville, Virginia